CLINICAL TRIAL: NCT05361707
Title: A Study to Evaluate the Efficacy and Safety of Tasimelteon in Treating Sleep Disturbances in Individuals With Autism Spectrum Disorder
Brief Title: Evaluating the Effects of Tasimelteon in Individuals With Autism Spectrum Disorder (ASD) and Sleep Disturbances
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VEC-162-3601
Record Dates: First submitted 2021-10-05; First posted 2022-05-05 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder; Sleep Disorder; Neurological Disorder; Sleep Disturbance
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Wake Disorders; Nervous System Diseases; Parasomnias

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tasimelteon (Experimental): Drug: Tasimelteon
  Interventions: Drug: Tasimelteon Oral Capsule, Tasimelteon Liquid Suspension

INTERVENTIONS:
Drug: Tasimelteon Oral Capsule, Tasimelteon Liquid Suspension — Once Daily

SUMMARY:
This is a multicenter, open-label study to evaluate the efficacy and safety of a daily single oral dose of tasimelteon in treating sleep disturbances in pediatric and adult participants with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written informed consent of the participant or legal guardian (and assent as required).
* A confirmed clinical diagnosis of Autism Spectrum Disorder (ASD) and a recent history of sleep disturbances.
* The sleep disturbance must not be a result of another diagnosable disorder or medication.
* Male or female between 2 and 65 years of age, inclusive.
* Willing and able to comply with study requirements and restrictions.

Exclusion Criteria:

* Inability to dose daily with tasimelteon or previous intolerance to tasimelteon.
* Indication of impaired liver function.
* Evidence of increased risk of self-harm.
* Pregnant or lactating females.
* A positive test for drugs of abuse.
* Other diagnosable causes of sleep disorders or use of medications that may cause sedation or stimulation.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in sleep time over the treatment period, as measured by sleep diary. | 12 weeks

SECONDARY OUTCOMES:
Improvement in objective sleep-wake parameters such as severity of condition, as measured by administered questionnaires. | 12 weeks
Improvement in objective behavioral parameters such as the participant's overall behavior, as measured by sleep diary in the Patient Global Impression of Severity Behavior Questionnaire (PGI-S Behavior). | 12 weeks
Assessment of safety and tolerability of daily single dose of tasimelteon, as measured by spontaneous reporting of adverse events (AEs). | 12 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Vanda Investigational Site, San Jose, California
  - Vanda Investigational Site, San Leandro, California
  - Vanda Investigational Site, Santa Monica, California
  - Vanda Investigational Site, Boulder, Colorado
  - Vanda Investigational Site, Staten Island, New York

IPD SHARING:
Plan to Share IPD: No